| Official Title: | A Multilevel Approach to Improving Colorectal Cancer |
|-----------------|-------------------------------------------------------|
| | Screening in Rural Communities of the FH/UW Catchment |
| | Area |
| NCT Number: | NCT05291988 |
| Document Type: | Informed Consent Form |
| Date of the | 6/14/2022 |
| Document: | |

#### Fred Hutchinson Cancer Center

# Informed Consent

# "Screen to Save" A Multilevel appraoch to improving colorectal cancer screening in rural communities of the FH/UW Catchment Area

Principal Investigator: Rachel M. Ceballos, PhD; Fred Hutchinson Cancer Center, 206-667-7806 Olympic Medical Center Research Contact: Tatyana Buzdnitskaya, RN, BSN, Nursing Research Coordinator, 360-582-2868

#### Important things to know about this study

You are invited to participate in this research study. Scientists at Fred Hutchinson Cancer Center and the Olympic Medical Cancer Center are working to learn more about providing colorectal cancer education and promote colorectal cancer screenings. Colorectal cancer screenings help to prevent the development of colorectal cancer.

If you agree to join the study you will be asked to complete a brief survey before and after the educational video.

You do not have to be in this study. And, you CAN receive a FIT Kit to have a colorectal cancer screening whether or not you participate in this project to tell us about the online education.

The following is a more complete description of this study.

# We would like you to join this research study

For this study, we are asking people to watch an online educational video and to complete two brief surveys, one before and one after watching the video about colorectal cancer.

If you agree to join the study,

- We will ask you to complete a brief questionnaire that will take about 5 minutes to complete.
   The questionnaire will ask basic questions about you (such as age and race/ethnicity, etc) and about your knowledge about colorectal cancer and interest in colorectal cancer screening.
- You will then watch the 9-minute video.
- The video will be followed by another brief questionnaire that will take an additional 5 minutes to complete. The questionnaire will ask about your colorectal cancer knowledge, your thoughts on the video, and your interest in colorectal cancer screening.

If you agree to join this study, we expect this will take no longer than 20 minutes to complete in total.

You do not have to join the study. You are free to say yes or no or to drop out after joining. There is no penalty or loss of benefits if you say no. Whatever you decide, your regular medical care will not change.

FHCRC IRB Approval JUN 14 2022 Document Released Date If you leave the study, your information cannot be removed from the study records.

#### What are the risks?

- While unlikely, the short questionnaire and video could cause you to feel uncomfortable a little stressed. Please note that you can skip any question you do not want to answer and that you are free to drop out of study at any time. There are no other risks known to you.
- There is a small risk of loss of confidentiality.

#### What are the benefits?

Although there are no benefits to those that join the study, the research could discover new ways to improve colorectal cancer education and, potentially, the number of people that are screened for colorectal cancer.

# Protecting your Privacy as an Individual and the Confidentiality of Your Personal Information

When studying your data, it will be **de-identified**. That is, we will remove your name, address or telephone number from the records. We will not share your data with other researchers or use it for any other reason outside of this study. However, some people or organizations may need to look at your research records for quality assurance or data analysis. They include:

- Researchers involved with this study at the Fred Hutchinson Cancer Center and the Olympic Medical Cancer Center.
- Institutional Review Boards (IRB), including the Fred Hutchinson Cancer Center IRB. An IRB is a group that reviews the study to protect your rights as a research participant.
- Office for Human Research Protections, and other agencies as required.

We will do our best to keep your personal information confidential. But we cannot guarantee total confidentiality. Your personal information may be given out if required by law. For example, a court may order study information to be disclosed. Such cases are rare.

We will not identify you or make your personal information available in any reports about this study, such as journal articles or presentations at scientific meetings. All study data will be presented without identifying individual participants in the study.

# Will you pay me to be in this study?

No payment will be made for completion of the study.

#### How much will this study cost me?

Participants will be responsible for their clinical care. All other components of the study are free of

charge.

#### What if you get sick or hurt after you join this study?

For a life-threatening problem, call 911 right away or seek help immediately. Contact your study doctor when the medical emergency is over or as soon as you can.

For all other medical problems or illness related to this research, immediately contact your primary care provider or healthcare team. They will treat you or refer you for treatment. You or your health insurance will have to pay for the treatment. There are no funds to pay you for a research-related injury, added medical costs, loss of a job, or other costs to you or your family. State or national law may give you rights to seek payment for some of these expenses. You do not waive any right to seek payment by signing this consent form.

Yor your insurer will be billed for treatment of problems or complications that result from your condition or from standard clinical care.

#### What will my information be used for?

Your information will be used for the purposes of this study.

#### Your rights

- You do not have to join this study. You are free to say yes or no.
- Although not anticipated, if you get sick or hurt in this study, you do not lose any of your legal rights to seek payment by signing this form.
- If you join this study, you do not have to stay in it. You may stop at any time (even before you start). There is no penalty for stopping. Your regular medical care would not change. You would have no penalty for stopping, but it would be better not to join the study if you think that you would change your mind later.

### Will my information and biological sample be used for future research?

Your information and tissue samples (even if made anonymous) will not be used for any research other than this study.

#### For more information

If you have questions or concerns about this study, you can talk to a member of the study team anytime.

| If you have questions about: | Call: |
|---|---|
| This study (including complaints and requests for information) | 206.667.7806, Dr. Rachel Ceballos, Fred Hutch, Associate Professor, Principal Investigator (PI) |
| | 360.582.2868, Tatyana Buzdnitskaya, RN, BSN, Olympic Medical Cancer Center, Nursing Research Coordinator |
| Your rights as a research participant | 206.667.5900 or email irodirector@fredhutch.org Director of Institutional Review Office, Fred Hutchinson Cancer Research Center |